CLINICAL TRIAL: NCT04659174
Title: An Open-label Extension Study to Assess the Long-term Safety, Tolerability, and Efficacy of KarXT in Subjects With DSM-5 Schizophrenia
Brief Title: An Extension Study to Assess Long-term Safety, Tolerability, and Efficacy of KarXT in Adult Patients With Schizophrenia (EMERGENT-4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAR-008
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — Oral xanomeline 50 mg/trospium chloride 20 mg BID on days 1-2 followed by xanomeline 100 mg/trospium chloride 20 mg BID on days 3-7. The dosage is increased to xanomeline 125 mg/trospium chloride 30 mg BID on days 8-364 unless the subject is experiencing adverse events from the xanomeline 100 mg/ trospium chloride 20 mg dose. Subjects who were increased to xanomeline 125 mg/trospium chloride 30 mg will have the option to return to xanomeline 100 mg/ trospium chloride 20 mg depending on clinical response and tolerability. Re-escalation to 125/30 BID or re-titration in cases in which the subject has been off KarXT for a longer period of time (at least a week) is allowed and will require a discussion between the principal investigator and the medical monitor.
  Other Names: KarXT

SUMMARY:
This is a Phase 3, multicenter, 53-week, outpatient, open-label extension (OLE) study to evaluate the long-term safety, tolerability, and efficacy of KarXT in subjects with Diagnostic and Statistical Manual-Fifth Edition (DSM-5) schizophrenia who previously completed the treatment period of one of the two Phase 3 double-blind studies, KAR-007 or KAR-009. In this OLE study, all subjects will receive KarXT (a fixed combination of xanomeline 125 mg and trospium chloride 30 mg twice daily [BID]) for up to 52 weeks regardless of treatment assignment in the preceding Phase 3 acute study. The primary objective of the study is to assess the long-term safety and tolerability of KarXT in subjects with a DSM-5 diagnosis of schizophrenia. The secondary objective of this study is to assess the long-term efficacy and monitor trough concentrations of xanomeline and trospium after administration of KarXT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 65 years, at time of enrollment into the preceding acute study (KAR-007/009).
2. Subject is capable of providing informed consent.

   1. A signed informed consent form must be provided before any study assessments are performed.
   2. Subject must be fluent in (oral and written) English (United States only) or local language (Ukraine only) to consent.
3. Subject has completed the treatment period on study drug (through Day 35 -2 days) of Studies KAR-007 or KAR-009.
4. Subject resides in a stable living situation, in the opinion of the investigator.
5. Subject has an identified, reliable informant/caregiver willing to be able to address some questions related to certain study visits, if needed. An informant/caregiver may not be necessary if the subject has been the patient of the investigator for ≥1 year.
6. Women of childbearing potential or men with sexual partners of childbearing potential must be sexually abstinent (in line with their preferred and usual lifestyle) or willing and able to use at least 1 highly effective method of contraception during the study and for at least 7 days after the last dose of KarXT. Sperm donation is not allowed for 7 days after the final dose of KarXT.

Exclusion Criteria:

1. Risk for suicidal behavior during the study as determined by the investigator's clinical assessment and Columbia-Suicide Severity Rating Scale (C-SSRS).
2. Any clinically significant abnormality, including any finding(s) from the physical examination, vital signs, ECG, or laboratory test at the end-of-treatment visit of Studies KAR-007 or KAR-009 that the investigator, in consultation with the medical monitor, would consider to jeopardize the safety of the subject.
3. Female subject is pregnant.
4. If, in the opinion of the investigator (and/or Sponsor), subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the investigator (and/or Sponsor), may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements.
5. Subjects with extreme concerns relating to global pandemics such as coronavirus disease 2019 (COVID-19) that preclude study participation.
6. Risk of violent or destructive behavior.
7. Subjects participating in another investigational drug or device trial or planning on participating in another clinical trial during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- United States (34):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - Advanced Research Center Inc, Bellflower, California
  - CITrials, Bellflower, California
  - Proscience Research Group, Culver City, California
  - Collaborative NeuroScience Research, LLC, Garden Grove, California
  - California Clinical Trial Medical Group, Glendale, California
  - Synergy San Diego, Lemon Grove, California
  - CNS Network, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - NRC Research Institute, Orange, California
  - California Neuropsychopharmacology Clinical Research Institute, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Collaborative Neuroscience Research, LLC., Torrance, California
  - Behavioral Clinical Research, Inc., Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Mitchell L. Glaser, Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - AMITA Health Center for Psychiatric Research, Hoffman Estates, Illinois
  - Pillar Clinical Research, Lincolnwood, Illinois
  - Arch Clinical Trials, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Community Clinical Research, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
- Ukraine (10):
  - Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council, Female Department #11, Male Department #12, Smila, Cherkasy Oblast
  - Dnipropetrovsk Regional Clinical Hospital named after I.I. Mechnikov, Dnipro
  - Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine, Kharkiv
  - Regional Clinical Psychiatric Hospital No. 3, Adult Psychiatric Department No. 3, Kharkiv
  - Kherson Regional Insititution of Mental Care of Kherson Regional Council Male Psychiatric Department #3, Femail Psychiatric Department #10, Kherson
  - Kyiv Regional Medical Incorporation "Psychiatry", Center for Novel Treatment and Rehabilitation of Psychotic Disorders, Kyiv
  - Lviv Regional Clinical Psychiatric Hospital, Department #20, Lviv
  - Lviv Regional Clinical Psychiatric Hospital, Department #25, Lviv
  - Regional Facility for Psychiatric Care of Poltava Regional Council, 2-A acute general psychiatric male ward, 5-B acute, quiet, general psychiatric female ward, Poltava State Medical University, Academic Department of Psychiatry, Addictology and Medical, Poltava
  - M.I. Pyrogov Vinnytsya National Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KarXT Arm A: Lead-in doses of KarXT (KarXT 50/20 BID). Dosing will be titrated to 100/20 BID on Days 3 to 7 and further titrated to 125/30 BID on Day 8, unless the participant continues to experience AE(s) from the previous dose increase of KarXT. All participants will have the option to return to KarXT 100/20 BID for the remainder of the treatment period. Participants received KarXT previously from KAR-007 and KAR-009.
- KarXT Arm B: Lead-in doses of KarXT (KarXT 50/20 BID). Dosing will be titrated to 100/20 BID on Days 3 to 7 and further titrated to 125/30 BID on Day 8, unless the participant continues to experience AE(s) from the previous dose increase of KarXT. All participants will have the option to return to KarXT 100/20 BID for the remainder of the treatment period. Participants received Placebo previously from KAR-007 and KAR-009.
Period: Overall Study
Arm/Group | KarXT Arm A | KarXT Arm B
Started (Started treatment) | 68 | 84
Completed (Completed treatment) | 19 | 16
Not Completed | 49 | 68
Not completed — Sponsor decision to discontinue study | 0 | 2
Not completed — Lost to Follow-up | 9 | 11
Not completed — Adverse Event | 8 | 5
Not completed — Withdrawal by Subject | 17 | 33
Not completed — Progressive disease | 0 | 2
Not completed — Other reasons | 0 | 2
Not completed — Participant fails to adhere to the protocol requirements | 14 | 9
Not completed — Alcohol or illegal drug use | 0 | 3
Not completed — Violation of entry criteria | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KarXT Arm A | KarXT Arm B | Total
Number analyzed (Participants) | 68 | 84 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (10.94) | 43.3 (12.07) | 44.9 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 48 | 66 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 64 | 76 | 140
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 47 | 93
  White | 21 | 35 | 56
  Other | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as events with an onset date on or after the first dose of KarXT. An Adverse Event is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at baseline, worsens during the study, regardless of the suspected cause of the event using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Time Frame: From first dose to end of study (Up to approximately 53 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 68 | 84
Participants | 36 | 45

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence, in the view of either the investigator or sponsor, that results in death; is life-threatening; results in inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity, and/or; is a congenital anomaly/birth defect using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Time Frame: From first dose to end of study (Up to approximately 53 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 68 | 84
Participants | 5 | 3

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) Leading to Study Drug Discontinuation
Description: as for outcome 1
Time Frame: From first dose to end of study (Up to approximately 53 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 68 | 84
Participants | 9 | 7

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 52
Description: The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function and the negative symptoms are the diminution or loss of normal functions. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms. Open-label Extension Baseline (OLEB) is defined as the most recent measurement prior to the first administration of study drug in KAR-008. The assessments performed on Visit 10 (Day 35) of studies KAR-007 or KAR-009 will be considered for OLEB baseline along with any additional procedures that will be performed on Day 0 of KAR-008.
Time Frame: Open-label extension baseline, week 52
Population: All participants who received at least 1 dose of KarXT and have a valid post-baseline PANSS assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 19 | 16
score on a scale | -9.0 (17.33) | -23.9 (22.06)

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Score at Week 52
Description: PANSS positive score is the sum of all PANSS 7 positive symptom scales with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe symptoms. Participants are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function such as hallucinations, delusions, grandiosity, and hostility. Open-label Extension Baseline (OLEB) is defined as the most recent measurement prior to the first administration of study drug in KAR-008. The assessments performed on Visit 10 (Day 35) of studies KAR-007 or KAR-009 will be considered for OLEB baseline along with any additional procedures that will be performed on Day 0 of KAR-008.
Time Frame: Open-labe extension baseline, week 52
Population: All participants who received at least 1 dose of KarXT and have a valid post-baseline PANSS assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 19 | 16
score on a scale | -3.2 (5.85) | -7.8 (6.38)

6. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Score at Week 52
Description: PANSS negative score is the sum of all PANSS 7 negative symptom scales with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe symptoms. Participants are rated from 1 to 7 on each symptom scale. The negative symptoms in schizophrenia are the diminution or loss of normal functions. Open-label Extension Baseline (OLEB) is defined as the most recent measurement prior to the first administration of study drug in KAR-008. The assessments performed on Visit 10 (Day 35) of studies KAR-007 or KAR-009 will be considered for OLEB baseline along with any additional procedures that will be performed on Day 0 of KAR-008.
Time Frame: Open-label extension baseline, week 52
Population: All participants who received at least 1 dose of KarXT and have a valid post-baseline PANSS assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 19 | 16
score on a scale | -2.1 (4.01) | -4.6 (5.06)

7. Secondary Outcome: Change From Baseline in PANSS Negative Marder Factor Score at Week 52
Description: PANSS Negative Marder Factor Score is the sum of 5 negative scales and 2 general scales (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance). Participants are rated from 1 to 7 on each symptom scale. Higher score indicates more severe symptoms. The negative symptoms in schizophrenia are the diminution or loss of normal functions. Open-label Extension Baseline (OLEB) is defined as the most recent measurement prior to the first administration of study drug in KAR-008. The assessments performed on Visit 10 (Day 35) of studies KAR-007 or KAR-009 will be considered for OLEB baseline along with any additional procedures that will be performed on Day 0 of KAR-008.
Time Frame: Open-label extension baseline, week 52
Population: All participants who received at least 1 dose of KarXT and have a valid post-baseline PANSS assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 19 | 16
score on a scale | -2.4 (4.22) | -5.1 (5.67)

8. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 52
Description: Completed independently by a clinician, the CGI-S categorizes the severity of the illness as: 1 = Normal, not at all ill; 2 = Borderline mentally ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; and 7 = Among the most extremely ill patients, by asking the clinical 1 question and providing a rating based upon observed and reported symptoms, behavior, and function in the past 7 days to reflect the average severity level across the 7 days. Higher score indicates more severe illness. Open-label Extension Baseline (OLEB) is defined as the most recent measurement prior to the first administration of study drug in KAR-008. The assessments performed on Visit 10 (Day 35) of studies KAR-007 or KAR-009 will be considered for OLEB baseline along with any additional procedures that will be performed on Day 0 of KAR-008.
Time Frame: Open-label extension baseline, week 52
Population: All participants who received at least 1 dose of KarXT and have a valid post-baseline CGI-S assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 19 | 16
score on a scale | -0.5 (1.12) | -1.2 (1.60)

9. Secondary Outcome: Percentage of PANSS Responders With >=30% Reduction in PANSS Total Score at Week 52
Description: A PANSS responder is defined as a participant with reduction from open-label extension baseline (OLEB) of at least a 30% improvement at Week 52 in the PANSS total score. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms. OLEB is defined as the most recent measurement prior to the first administration of study drug in KAR-008. The assessments performed on Visit 10 (Day 35) of studies KAR-007 or KAR-009 will be considered for OLEB baseline along with any additional procedures that will be performed on Day 0 of KAR-008.
Time Frame: At week 52
Population: All participants who received at least 1 dose of KarXT and have a valid post-baseline PANSS assessment
Measure: Number; unit: Percentage of participants
Arm/Group | KarXT Arm A | KarXT Arm B
Number analyzed (Participants) | 19 | 16
Percentage of participants | 42.1 | 56.3

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events from the date of first dose until study completion (Up to approximately 53 weeks).
Description: All participants who received at least one dose of study treatment.
Arm/Group | KarXT Arm A | KarXT Arm B
All-Cause Mortality (participants affected / at risk) | 0/68 | 1/84
Serious Adverse Events (participants affected / at risk) | 5/68 | 3/84
Other Adverse Events (participants affected / at risk) | 19/68 | 31/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT Arm A (N=68) | KarXT Arm B (N=84)
Death (General disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT Arm A (N=68) | KarXT Arm B (N=84)
Constipation (Gastrointestinal disorders) | 4 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 6 | 8
Vomiting (Gastrointestinal disorders) | 2 | 11
Weight increased (Investigations) | 3 | 6
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT04659174/Prot_SAP_000.pdf